CLINICAL TRIAL: NCT05861219
Title: Alternative Haemodiafiltration in Summer Season for Chronic Kidney Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MANAR SALAH AHMED BARAKAT, assisstant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: alternative HDF in CKD
Record Dates: First submitted 2023-04-27; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Sweating

STUDY DESIGN:
Intervention Model Description: Chronic kidney disease stage 3,4
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chronic kidney disease patients stage 3 and 4 (Experimental): 50 chronic kidney disease patients stage 3 and 4 will perform mild exercise and water immersion
  Interventions: Behavioral: water immersion

INTERVENTIONS:
Behavioral: water immersion — mild physical activity then water immersion in tub

SUMMARY:
Hemodiafiltration is a renal replacement technique combining diffusion and convection to enhance solute removal. Post dialyser replacement fluid is administered to achieve the target fluid balance. The skin is the largest human organ playing an important role in thermal and Na regulation and skin blood flow is 8.5-10%of cardiac output .

DETAILED DESCRIPTION:
Sweat contains electrolytes, creatinine and urea, with higher excretion by mild physical exercise. These findings motivate studies investigating the effect of stimulated sweating on volume control in kidney disease patients. Using sweat as the vehicle for removing molecules normally excreted in the urine was identified some decades ago. sweat urea concentration could reach 5.5 to 50 times the serum concentration .

Physical inactivity was reported as the fourth leading cause of death from chronic disease worldwide. Warm water immersion (37-46◦C) increases limb blood flow, and muscle heating activates regulators of mitochondrial biogenesis. water immersion represent diffusion .the average person sweats between (0.8- 1.4) liters during an hour of exercise, drinking water represent water replacement .

Particularly, urea concentrations in sweat are persistently elevated in uremic patients. The 24-hour urinary urea excretion in summer was 1/4 the quantity in winter in uremic patients, indicating the compensatory urea excretion in sweat gland fluid . Sweat glands are inactive except above 29°C, due to a concentration gradient within the stratum corneum, results in continuous water convection from within the body through the skin and into the environment.

In our study we stimulate sweating of chronic kidney disease patients through mild physical activity as walking then they immersied in water to enhance waste excretion through skin.Evaluation of these patients will be done through following up blood pressure,laboratory investigations as kidney function test sodium, potassium,phosphorus levels and uric acid.

ELIGIBILITY:
Inclusion Criteria:

chronic kidney disease group:

1. stage 3,4
2. Age(18-60)yrs old.
3. Not on dialysis.
4. Without uremic symptoms nor standard indication for dialysis

Exclusion Criteria:

1. History of cerebrovascular accidents.
2. History of advanced cardiac disease (heart failure, recent acute coronary syndrome, and cardiac arrhythmia).
3. Active skin lesion
4. volume overload. 5- advanced liver cirrhosis, respiratory failure, and malignancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-21 (Estimated); Primary Completion 2024-06-21 (Estimated); Study Completion 2025-06-21 (Estimated)

PRIMARY OUTCOMES:
assessment of improvement of kidney function test( urea and creatinine) | 1 year
  kidney function test (serum urea and creatinine im mg\dl) will measured before the procedure with weekly follow up
assess improvement of blood pressure | 1 year
  follow up blood pressure (systolic and diastolic blood pressure in mm hg)

SECONDARY OUTCOMES:
assessment of improvement in serum potassium level | 1 year
  measure potassium level in mmol\L with weekly follow up

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Elshazly, professor, Study Chair — professor

IPD SHARING:
Plan to Share IPD: Yes
study design results
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 to 3 years

REFERENCES:
- [Background] Ronco C. Hemodiafiltration: Technical and Clinical Issues. Blood Purif. 2015;40 Suppl 1:2-11. doi: 10.1159/000437403. Epub 2015 Sep 8. PMID 26344507
- [Background] Baker LB. Physiology of sweat gland function: The roles of sweating and sweat composition in human health. Temperature (Austin). 2019 Jul 17;6(3):211-259. doi: 10.1080/23328940.2019.1632145. eCollection 2019. PMID 31608304
- [Background] Huang CT, Chen ML, Huang LL, Mao IF. Uric acid and urea in human sweat. Chin J Physiol. 2002 Sep 30;45(3):109-15. PMID 12817713
- [Background] Blank IH, Moloney J 3rd, Emslie AG, Simon I, Apt C. The diffusion of water across the stratum corneum as a function of its water content. J Invest Dermatol. 1984 Feb;82(2):188-94. doi: 10.1111/1523-1747.ep12259835. PMID 6693781
- [Background] Joo CH, Allan R, Drust B, Close GL, Jeong TS, Bartlett JD, Mawhinney C, Louhelainen J, Morton JP, Gregson W. Passive and post-exercise cold-water immersion augments PGC-1alpha and VEGF expression in human skeletal muscle. Eur J Appl Physiol. 2016 Dec;116(11-12):2315-2326. doi: 10.1007/s00421-016-3480-1. Epub 2016 Oct 3. PMID 27699485
- [Background] al-Tamer YY, Hadi EA, al-Badrani II. Sweat urea, uric acid and creatinine concentrations in uraemic patients. Urol Res. 1997;25(5):337-40. doi: 10.1007/BF01294662. PMID 9373914